CLINICAL TRIAL: NCT00384384
Title: Glycyrrhetinic Acid-Effect on Serum Potassium and Insulin Resistance in Dialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: S51/05
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: End Stage Renal Disease
Keywords: Dialysis; Serum potassium; 18b glycyrrhetinic acid; insulin sensitivity
MeSH Terms: conditions — Kidney Failure, Chronic; Insulin Resistance

INTERVENTIONS:
Drug: oral 18B Glycyrrhetinic acid versus placebo

SUMMARY:
Background: 18B Glycyrrhetinic acid (active compound of Licorice) decreases serum potassium via enhanced renal potassium loss in healthy individuals and thereby inducing renal sodium retention and arterial hypertension.In dialysis patients this mechanism is disturbed and compensatory intestinal potassium secretion is enhanced. 18B Glycyrrhetinic acid is an inhibitor of 11B Hydroxysteroid dehydrogenase type 1 (11b HSD1). Inhibition of 11 b HSD1 offers a novel potential therapy to lower intracellular cortisol concentrations and thereby enhance insulin sensitivity.

Hypothesis: Glycyrrhetinic acid decreases serum potassium by enhanced intestinal excretion in dialysis patients and increases insulin sensivity by inhibition of 11b HSD

Methods: double blind, 6 month cross over trial comparing oral 18b Glycyrrhetinic acid with placebo in 24 nondiabetic dialysis patients.

Endpoints: predialytic serum potassium levels, insuline sensitivity assessed by fasting glucose and fasting insulin concentrations

ELIGIBILITY:
Inclusion Criteria:

* dialysis patients (>3 months)

Exclusion Criteria:

* diabetics
* hospital stay in the last 4 weeks

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Start 2006-08; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felix J Frey, Prof, Principal Investigator — Department of Nephrology and Hypertension, University hospital of Berne
Locations (1):
- Department of nephrology and hypertension, University hospital of berne, Bern, Switzerland

REFERENCES:
- [Derived] Farese S, Kruse A, Pasch A, Dick B, Frey BM, Uehlinger DE, Frey FJ. Glycyrrhetinic acid food supplementation lowers serum potassium concentration in chronic hemodialysis patients. Kidney Int. 2009 Oct;76(8):877-84. doi: 10.1038/ki.2009.269. Epub 2009 Jul 29. PMID 19641483